CLINICAL TRIAL: NCT01202812
Title: Phase II Randomized Double-Blind Placebo-Controlled Trial of the Omega-3 Fatty Acids Eicosapentaenoic (EPA) and Docosahexaenoic Acid (DHA) in Pediatric Sickle Cell Disease (SCD)
Brief Title: A Randomized Trial of LOVAZA in Pediatric Sickle Cell Disease (SCD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Drexel University (Other); GlaxoSmithKline (Industry)
Responsible Party: Marie Stuart, MD, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10F.161
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Sickle Cell Disease; HEMOGLOBIN SS; Hemoglobin S Beta-0 Thalassemia; Inflammation; Quality of Life
Keywords: Sickle Cell Anemia; Sickle Cell Disease; Hemoglobin SS Disease; Hemoglobin S beta-0 Thalassemia; Inflammation; Quality of Life; Sickle Thalassemia; C-Reative Protein; Hemolytic Anemia; Hemostasis; Biomarkers; Coagulation; Omega-3 Fatty Acids; Eicosapentaenoic Acid; Docosahexaenoic Acid; Fish Oils; Drug: Placebo; Drug: LOVAZA
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation; Anemia, Hemolytic; Thrombosis | interventions — Docosahexaenoic Acids; Fish Oils; Eicosapentaenoic Acid; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOVAZA (Experimental)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids: Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA)
- Placebo capsule (Placebo Comparator)
  Interventions: Other: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids: Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) — Eicosapentaenoic Acid (EPA)/Docosahexaenoic Acid (DHA) 30mg/kg (LOVAZA capsules) given by mouth daily for 6 months.
  Other Names: - Fish Oils; - Eicosapentaenoic Acid; - Docosahexaenoic Acid; - Omega-3 Fatty Acid
  Arms: LOVAZA
Other: Placebo Capsules — Placebo capsules given by mouth daily for 6 months.
  Other Names: - Placebo
  Arms: Placebo capsule

SUMMARY:
The purpose of the study is to determine the effectiveness of LOVAZA (fish oil capsules) to decrease inflammation in children and adolescents with Sickle Cell Disease (SCD). It has been found that besides the damage caused by sickle red blood cells themselves, the inflammatory response that occurs in SCD patients could potentially play a significant role in the occurrence of painful episodes or pain crises. The investigators will also study whether the subject/caregiver feels that there is an improvement in the child's quality of life by taking the medication. Besides the effect of LOVAZA on inflammation,the investigators are also testing whether the drug will have a beneficial effect on blood clotting ability (which is known to be increased in SCD) and on the anemia (low red blood cells) that is part of the disease entity.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible for enrollment into the study:

* Participant has signed the informed consent/assent with parent signing informed consent as age appropriate.
* Established diagnosis of HbSS or HbSβo Thal.
* History of ≥3 vasocclusive pain events in preceding 12 months.
* Regular compliance with comprehensive care.
* Aged 10 years or greater and less than 20 years.
* At enrollment, subject should be in his/her steady or baseline state.

Exclusion Criteria

* Subjects with Hb levels <5.5gm/dL.
* Inability to take or tolerate oral medications.
* Poor compliance with previous treatment regimens.
* Hepatic dysfunction (SGPT also known as ALT >2X upper limit of normal or conjugated bilirubin >2X the patients baseline within the last 6 weeks).
* Renal dysfunction (A creatinine level within the past 6 weeks of ≥ 1.0mg/dL for children and ≥ 1.2mg/dL for a subject ≥ 18 years of age).
* Allergy to fish or shell fish.
* Triglyceride levels <80mg/dL.
* Pregnancy.
* Chronic Transfusion Therapy.
* Transfusion within the last 30 days.
* Persistent pain from sickle-complications (e.g. avascular necrosis).
* A vasocclusive pain episode lasting longer than 2 weeks or >12 pain episodes in preceding year.
* Daily narcotic usage.
* Treatment with any investigational drug or regular fish oil supplementations in last 60 days.
* Currently receiving another investigational agent, or on such an agent with the last 60 days.
* Dosage changes in preceding 3 months if on hydroxyurea.
* Bleeding disorder or patient on concomitant anti-coagulation.
* Conditional or abnormal TCD result or stroke.
* Other chronic illness that could adversely affect subjects performance such as HIV or TB.
* Children in Care (CiC): A child in care is a child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
To determine whether supplementation with LOVAZA will exert an anti-inflammatory effect by decreasing levels of the inflammatory biomarker high sensitivity C Reactive Protein (hsCRP) in children and adolescents with Sickle Cell Disease (SCD). | 6 months

SECONDARY OUTCOMES:
To determine whether supplementation with LOVAZA will increase health-associated quality of life (QoL) responses as they relate to clinical vasocclusive events (VOC) in children and adolescents with Sickle Cell Disease (SCD). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Stuart, M.D., Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Drexel University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Tomer A, Kasey S, Connor WE, Clark S, Harker LA, Eckman JR. Reduction of pain episodes and prothrombotic activity in sickle cell disease by dietary n-3 fatty acids. Thromb Haemost. 2001 Jun;85(6):966-74. PMID 11434703
- [Background] Krishnan S, Setty Y, Betal SG, Vijender V, Rao K, Dampier C, Stuart M. Increased levels of the inflammatory biomarker C-reactive protein at baseline are associated with childhood sickle cell vasocclusive crises. Br J Haematol. 2010 Mar;148(5):797-804. doi: 10.1111/j.1365-2141.2009.08013.x. Epub 2009 Dec 8. PMID 19995398
- [Background] Dampier C, Lieff S, LeBeau P, Rhee S, McMurray M, Rogers Z, Smith-Whitley K, Wang W; Comprehensive Sickle Cell Centers (CSCC) Clinical Trial Consortium (CTC). Health-related quality of life in children with sickle cell disease: a report from the Comprehensive Sickle Cell Centers Clinical Trial Consortium. Pediatr Blood Cancer. 2010 Sep;55(3):485-94. doi: 10.1002/pbc.22497. PMID 20658620
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255